CLINICAL TRIAL: NCT02911701
Title: Effect of Acetaminophen on Postpartum Blood Pressure Control in Preeclampsia With Severe Features
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Luis Izquierdo, Associate Professor of Clinician Education, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16-147
Record Dates: First submitted 2016-09-09; First posted 2016-09-22 (Estimated); Results first posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Pre-Eclampsia; HELLP Syndrome; Eclampsia
MeSH Terms: conditions — Pre-Eclampsia; HELLP Syndrome; Eclampsia | interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acetaminophen (Experimental): Study participants randomized to the acetaminophen group will receive 650mg of acetaminophen orally every 6 hours during their postpartum hospital stay.
  Interventions: Drug: Acetaminophen
- Ibuprofen (Active Comparator): Study participants randomized to the ibuprofen group will receive 600mg of ibuprofen orally every 6 hours during their postpartum hospital stay.
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Acetaminophen
  Other Names: Tylenol
  Arms: Acetaminophen
Drug: Ibuprofen
  Other Names: Motrin
  Arms: Ibuprofen

SUMMARY:
NSAIDs, specifically cyclo-oxygenase (COX) inhibitors, are known to increase blood pressure over time in non-pregnant adults, but the effect of COX-inhibitors on blood pressure in the setting of preeclampsia have not been well studied. This study aims to assess the effect of avoiding COX-inhibitors on postpartum blood pressure control among women diagnosed with preeclampsia with severe features. Eligible women will be randomized to receive either acetaminophen or ibuprofen for postpartum pain control. Both agents are first line therapies for pain control although ibuprofen has better pain control than acetaminophen. The primary outcome will be duration of postpartum severe-range hypertension.

DETAILED DESCRIPTION:
The proposed study is a randomized, controlled, double-masked trial comparing the effect of postpartum acetaminophen and ibuprofen on blood pressure among women with preeclampsia. Study participants will be randomized to receive either acetaminophen or ibuprofen for mild postpartum pain control. Study participants, study personnel and providers will be blinded to randomization status of study participants.

Potential study participants will be enrolled when they are diagnosed with a severe hypertensive disorder of pregnancy. This will usually occur prior to delivery, but may occur up to 6 hours after delivery. Patients diagnosed with preeclampsia without severe features will also be approached and enrolled at the time of diagnosis in anticipation for possible progression to preeclampsia with severe features. Once enrolled, study participants will not be randomized until delivery, at which time they will be randomized to receive either acetaminophen or ibuprofen for mild postpartum pain. Both groups will have available oxycodone for moderate to severe pain, per our routine. Study group allocation will only be known by the investigational pharmacy. The ibuprofen and acetaminophen will be made to appear identical to each other and will be unmarked through encapsulation. Block randomization will be used to ensure equal allocation to the two study arms.

For the duration of study participation, study participants will undergo postpartum monitoring with vital sign measurements (including blood pressure) every 4 hours, pain assessment with each administration of study medication, as well as daily evaluation of laboratory studies until they have normalized to the satisfaction of their provider. Study participants will receive the study drug every 6 hours from the time of delivery until hospital discharge, unless they refuse. Study participation will be complete upon hospital discharge. Study participants will be contacted by a study team member 6 weeks after delivery to ask about any additional complications or symptoms requiring visits to the emergency department or hospital readmission. Descriptive factors and clinical outcomes will be extracted from the medical record and de-identified by study personnel during each day of study participation.

ELIGIBILITY:
Inclusion Criteria:

* ability to give informed consent
* diagnosis of a "severe" hypertensive disorder of pregnancy:
* preeclampsia with severe features
* chronic hypertension with superimposed preeclampsia with severe features
* HELLP syndrome: hemolysis, elevated liver function tests, low platelets
* eclampsia
* not yet delivered or less than 6 hours after delivery

Exclusion Criteria:

* current incarceration
* serum creatinine > 1.0 mg/dL or suspicion of acute kidney injury
* AST (aspartate aminotransferase) >200 unit/L
* ALT (alanine aminotransferase) > 200 unit/L
* known allergy or sensitivity to NSAIDs or acetaminophen
* delivery > 6 hours prior to enrollment
* chronic kidney disease
* chronic liver disease
* prior liver transplant
* chronic infectious hepatitis
* gastritis
* gastro-esophageal reflux disease (GERD)
* peptic ulcer disease
* bleeding disorder
* provider feels that participation is not in the best interest of the patient

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-09; Primary Completion 2017-11-07 (Actual); Study Completion 2018-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luis Izquierdo, MD, MBA, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico Health Sciences Center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Acetaminophen: Study participants randomized to the acetaminophen group will receive 650mg of acetaminophen orally every 6 hours during their postpartum hospital stay.
  Acetaminophen
- Ibuprofen: Study participants randomized to the ibuprofen group will receive 600mg of ibuprofen orally every 6 hours during their postpartum hospital stay.
  Ibuprofen
Period: Overall Study
Arm/Group | Acetaminophen | Ibuprofen
Started | 50 | 50
Completed | 47 | 46
Not Completed | 3 | 4
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acetaminophen | Ibuprofen | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.5 (6.4) | 31.9 (5.9) | 31.2 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 50 | 100
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ethnicity: Hispanic | 20 | 20 | 40
  Race/ethnicity: White | 13 | 11 | 24
  Race/ethnicity: Black | 1 | 2 | 3
  Race/ethnicity: Asian | 0 | 2 | 2
  Race/ethnicity: Native American | 12 | 9 | 21
  Race/ethnicity: Other | 4 | 6 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50 | 50 | 100
mode of delivery [Count of Participants; unit: Participants]
  Vaginal | 32 | 25 | 57
  Operative vaginal | 1 | 1 | 2
  Cesarean | 17 | 24 | 41
Parity [Count of Participants; unit: Participants]
  Nulliparous | 19 | 18 | 37
  Multiparous | 31 | 32 | 63
chronic hypertension requiring treatment [Count of Participants; unit: Participants] | 7 | 8 | 15
need for IV Antihypertensives before delivery [Count of Participants; unit: Participants] | 37 | 42 | 79

OUTCOME MEASURES:

1. Primary Outcome: Duration of Severe-range Hypertension After Delivery
Description: length of time from delivery to the last severe range blood pressure (160/110mm Hg) measured
Time Frame: duration of postpartum hospitalization (approximately 3-7 days)
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | Acetaminophen | Ibuprofen
Number analyzed (Participants) | 50 | 50
hours | 38.0 [29.4 to 51.3] | 35.3 [27.2 to 47.5]
Statistical Analysis 1: Comparison: Acetaminophen vs Ibuprofen; Test type: Superiority; p = 0.3, maxim

2. Secondary Outcome: Length of Hospitalization
Description: number of days from delivery until hospital discharge
Time Frame: duration of postpartum hospitalization (approximately 3-7 days)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Acetaminophen | Ibuprofen
Number analyzed (Participants) | 50 | 50
days | 4.0 (1.3) | 3.8 (1.4)

3. Secondary Outcome: Mean Arterial Pressure Over the Entire Postpartum Hospitalization
Description: computed mean arterial pressure using all measured blood pressures during postpartum hospitalization
Time Frame: duration of postpartum hospitalization (approximately 3-7 days)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Acetaminophen | Ibuprofen
Number analyzed (Participants) | 50 | 50
mmHg | 97.3 (9.1) | 37.6 (6.2)

4. Secondary Outcome: Mean Arterial Pressure, Stratified by Postpartum Day 1, 2, 3, Etc.
Description: computed mean arterial pressure using all measured blood pressures during postpartum hospitalization, stratified by postpartum day (1, 2, 3, etc.)
Time Frame: duration of postpartum hospitalization (approximately 3-7 days)
Population: Data not collected
Arm/Group | Acetaminophen | Ibuprofen
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Mean Total Number of Severe Range Blood Pressure Measurements in Each Study Arm.
Description: mean total number of severe range blood pressure (defined as SBP >160mmGh or DBP >110mmHg) measurements in each study arm
Time Frame: duration of postpartum hospitalization (approximately 3-7 days)
Population: Data not collected
Arm/Group | Acetaminophen | Ibuprofen
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Proportion of Study Participants in Each Study Arm Who Have Any Postpartum Severe Range BPs
Description: Severe-range hypertension (defined as SBP > 160 mmHg or DBP >1100 mmHg) during postpartum stay
Time Frame: duration of postpartum hospitalization (approximately 3-7 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Acetaminophen | Ibuprofen
Number analyzed (Participants) | 50 | 50
Participants | 31 | 34

7. Secondary Outcome: Mean Maximum Measured Blood Pressure for Entire Postpartum Hospitalization (in mm Hg)
Time Frame: duration of postpartum hospitalization (approximately 3-7 days)
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Acetaminophen | Ibuprofen
Number analyzed (Participants) | 50 | 50
mm Hg | 165 (15) | 168 (16)

8. Secondary Outcome: Proportion of Study Participants Requiring the Use of Scheduled Oral Antihypertensives at Discharge
Time Frame: duration of postpartum hospitalization (approximately 3-7 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Acetaminophen | Ibuprofen
Number analyzed (Participants) | 50 | 50
Participants | 31 | 33

9. Secondary Outcome: Number of Scheduled Oral Antihypertensive Agents Required at Discharge
Time Frame: duration of postpartum hospitalization (approximately 3-7 days)
Population: Data not collected
Arm/Group | Acetaminophen | Ibuprofen
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Need for Antihypertensives (Either Oral or Intravenous) for Acute Lowering of Blood Pressure
Description: Proportion in each arm who required one or more doses of antihypertensive medication given for acute lowering of BP
Time Frame: duration of postpartum hospitalization (approximately 3-7 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Acetaminophen | Ibuprofen
Number analyzed (Participants) | 50 | 50
Participants | 26 | 30

11. Secondary Outcome: The Proportion of Study Participants Requiring the Use of Intravenous Antihypertensives
Description: The proportion of study participants in each study arm who require any IV antihypertensives to acutely lower blood pressure during their postpartum hospital stay.
Time Frame: duration of postpartum hospitalization (approximately 3-7 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Acetaminophen | Ibuprofen
Number analyzed (Participants) | 50 | 50
Participants | 26 | 30

12. Secondary Outcome: Mean Daily Pain Level, as Reported by Patient on Scale From 1-10, Stratified by Postpartum Day
Description: Mean daily pain level, as reported by patient on scale from 1-10 (10 is most severe).
Time Frame: duration of postpartum hospitalization (approximately 3-7 days)
Population: Clinical ascertainment of pain level was of low quality and so was not analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acetaminophen | Ibuprofen
Number analyzed (Participants) | 47 | 44
units on a scale | 2.4 (2.3) | 1.8 (1.7)

13. Secondary Outcome: Use of Opioid Analgesics, Measured in Morphine Milligram Equivalents Per Day, Stratified by Postpartum Day
Time Frame: duration of postpartum hospitalization (approximately 3-7 days)
Measure: Mean (Standard Deviation); unit: morphine equivalents, mg
Arm/Group | Acetaminophen | Ibuprofen
Number analyzed (Participants) | 50 | 50
morphine equivalents, mg
  postpartum day 0 | 22.6 (13.9) | 22.1 (25.1)
  postpartum day 1 | 32.3 (30) | 27.5 (18.7)
  postpartum day 2 | 45.4 (32.3) | 28.9 (18.9)

14. Secondary Outcome: Serum Creatinine Trend From Day of Delivery to Day of Discharge
Time Frame: duration of postpartum hospitalization (approximately 3-7 days)
Population: data not collected
Arm/Group | Acetaminophen | Ibuprofen
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Mean Drop in Hematocrit From Pre-delivery to the Nadir Prior to Discharge
Description: Mean difference in hematocrit from pre-delivery to postpartum nadir prior to discharge
Time Frame: duration of postpartum hospitalization (approximately 3-7 days)
Population: Data not collected
Arm/Group | Acetaminophen | Ibuprofen
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Composite of Adverse Events
Description: Adverse events include seizure, stroke, posterior reversible encephalopathy syndrome, repeat course of IV magnesium sulfate for seizure prophylaxis.
Time Frame: duration of postpartum hospitalization (approximately 3-7 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Acetaminophen | Ibuprofen
Number analyzed (Participants) | 50 | 50
Participants | 0 | 0

17. Secondary Outcome: Proportion of Study Participants in Each Study Arm With New Onset Postpartum Elevation of Liver Function Tests (AST, ALT) Above Twice the Normal Limit
Description: AST: Aspartate aminotransferase; ALT: alanine aminotransferase
Time Frame: duration of postpartum hospitalization (approximately 3-7 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Acetaminophen | Ibuprofen
Number analyzed (Participants) | 50 | 50
Participants | 1 | 0

18. Secondary Outcome: Proportion of Study Participants in Each Study Arm With New Onset Postpartum Acute Kidney Injury
Description: Acute kidney injury is defined as serum creatinine > 1.1mg/dL or double the baseline value
Time Frame: duration of postpartum hospitalization (approximately 3-7 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Acetaminophen | Ibuprofen
Number analyzed (Participants) | 50 | 50
Participants | 0 | 0

19. Secondary Outcome: Proportion of Study Participants in Each Study Arm With Delayed Postpartum Hemorrhage
Description: Delayed postpartum hemorrhage is defined as > 1000 mL of blood loss occuring > 24 hours after delivery
Time Frame: duration of postpartum hospitalization (approximately 3-7 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Acetaminophen | Ibuprofen
Number analyzed (Participants) | 50 | 50
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Duration of postpartum hospitalization, up to 2 weeks
Arm/Group | Acetaminophen | Ibuprofen
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 1/50 | 3/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acetaminophen (N=50) | Ibuprofen (N=50)
Inpatient readmission (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 3 (3) — exacerbation of preeclampsia requiring readmission
Acute postpartum elevation of liver function tests (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-17): https://cdn.clinicaltrials.gov/large-docs/01/NCT02911701/Prot_SAP_000.pdf